CLINICAL TRIAL: NCT03884582
Title: Observational Study to Detect Cough and Wheeze Sounds Using the CoVa Monitoring System 3
Brief Title: Observational Study Using the CoVa Monitoring System 3
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: RMD-IRB-0001
Record Dates: First submitted 2019-03-17; First posted 2019-03-21 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HealthyVolunteers
  Interventions: Device: Cova Monitoring System 3

INTERVENTIONS:
Device: Cova Monitoring System 3 — Healthy Volunteers

SUMMARY:
Asthma is a complex and chronic inflammatory disorder which is associated with reversible airway obstruction and bronchial hyperresponsiveness. It is one of the most prevalent chronic diseases in children and prevalence further increases worldwide. Typical symptoms of asthma are breathlessness, cough, wheezing and chest tightness. These symptoms are particularly prevalent at night-time. Understanding and tracking these symptoms can lead to better management of asthma.

Auscultation using a stethoscope is standard clinical practice, however there is currently no available solution to detect respiratory sounds throughout the day and night.

The aim of this study is to investigate the feasibility of detecting respiratory sounds in healthy children with the CoVa patch.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between the ages of 4 - 17 years old at the time of consent
* Participant and/or family member/carer willing to give written consent
* Participant and/or family member/carer who can read and comprehend english

Exclusion Criteria:

* Subject believed to be unsuitable for inclusion by the Principle Investigator
* Subject is pregnant at time of consent
* Subject is currently enrolled in another medical study

Ages: 4 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Ability to detect simulated respiratory sounds including coughing and wheezing or identify subjects which have asthma related respiratory issues | 2 Weeks
  Subjects will be asked to simulate coughing and wheezing sounds. This data will be analyzed by using a phonocardiogram (microphone) sensor.

SECONDARY OUTCOMES:
Ability to detect simulated respiratory sounds including wheeze and cough during movement such a simulated situation of moving in bed. | 2 Weeks
  Subjects will be asked to simulate coughing and wheezing sounds. This data will be analyzed by using a phonocardiogram (microphone) sensor while the subject is moving in the bed.

CONTACTS AND LOCATIONS:
Locations (1):
- toSense,Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No